CLINICAL TRIAL: NCT03692962
Title: Linking the Change in Decision-making After Sleep Restriction to the Restorative Function of Sleep
Brief Title: Decision-making After Sleep Restriction
Acronym: DM-SR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Baumann (Other)
Collaborators: Swiss Federal Institute of Technology in Zurich (ETH Zurich) (Unknown)
Responsible Party: Sponsor-Investigator, Christian Baumann, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DM-SR
Record Dates: First submitted 2018-06-04; First posted 2018-10-02 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Sleep Restriction
MeSH Terms: interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep restriction without acoustic stimulation (Sham Comparator)
  Interventions: Behavioral: Sleep restriction
- Sleep restriction with acoustic stimulation (Experimental)
  Interventions: Behavioral: Sleep restriction; Other: Acoustic stimulation

INTERVENTIONS:
Behavioral: Sleep restriction — Time in bed will be restricted to 5 hours per night for 7 nights.
Other: Acoustic stimulation — Brief tones will be presented time-locked to ongoing slow waves during deep sleep.
  Arms: Sleep restriction with acoustic stimulation

SUMMARY:
The aim of this project is to investigate whether enhancing sleep intensity locally in the prefrontal cortex (PFC) can counteract a deterioration of cognitive control and therefore the previously described increase in risk seeking during chronic sleep restriction. To this end, a controlled, counter-balanced study, consisting of two weeks of sleep restriction will be performed. During one of the sleep restriction weeks, sleep intensity in the PFC will be non-invasively enhanced by acoustic stimulation of slow waves during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-21 years or 26-30 years,
* Right-handedness,
* Good general health,
* Good understanding of German language (as all information is provided in German)
* Signed Informed Consent after being informed.

Exclusion Criteria:

* Contraindications on ethical grounds,
* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc),
* Known or suspected non-compliance, drug or alcohol abuse (> 5dl wine/ >1l beer daily),
* Regular medication intake,
* Enrolment into a clinical trial within last 4 weeks,
* Diseases or lesions of the nervous system (acute or residual included neurological and psychiatric diseases),
* Sleep disorders (e.g. Insomnia, sleep apnoea, restless leg syndrome, narcolepsy, etc.),
* Sleep complaints in general or excessive daytime sleepiness (Pittsburgh Sleep Quality Index > 5; Epworth Sleepiness Scale ≥ 11),
* Irregular sleep-wake rhythm (e.g. shift working),
* Long (> 10 hours per night) or short sleepers (< 7 hours per night),
* Sleep efficiency < 80% in screening night,
* Travelling with time lag less than 1 month ago (or planning to do so within 1 month prior to or during the study),
* > 5 drinks or food items containing caffeine per day,
* > 5 cigarettes per day,
* Body Mass Index < 19 or > 30 kg/m2,
* Skin allergy or very sensitive skin
* Student of one of the following subjects: Mathematics, Physics, Computer Science, Economics, or Psychology (since students of these subjects have profound knowledge of probability calculations, which could interfere with our measurements in decision-making).
* Red-Green Colour-Blindness (as the Risk Task requires the distinction between red and green),
* History of claustrophobia,
* Known hearing disorder (as acoustic stimuli will be applied during sleep),
* Magnetic Resonance (MR) contraindication (such as pacemaker, implanted pumps, shrapnel, etc.; full MR Screening form will be filled out).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
risk-premium | comparison of change from baseline after 7 nights of sleep restriction with acoustic stimulation to change from baseline after 7 nights of sleep restriction without acoustic stimulation
  risk-preference (i.e. risk premium assessed with the risk Task as described in Maric et al. 2017 Ann Neurol) after chronic sleep restriction with and without acoustic Stimulation will be quantified by the risk-premium derived from the choices made in the risk-task as described in Maric et al. 2017 Ann Neurol.

SECONDARY OUTCOMES:
high-density electroencephalography (hdEEG) marker of sleep pressure | assessed during first and last sleep restriction nights in comparison to baseline values
  Slow wave activity (SWA) assessed by hd-EEG with 128 electrodes
brain metabolites | before to after 7 nights of sleep restriction with and without acoustic stimulation
  Glutamate and gamma-aminobutyric acid (GABA) concentration in the right prefrontal Cortex assessed by magnetic resonance (MR) spectroscopy
vigilance measures | before to after 7 nights of sleep restriction with and without acoustic stimulation
  Performance impairments in the psychomotor-vigilance task
deception willingness | before to after 7 nights of sleep restriction with and without acoustic stimulation
  deception willingness measured by the willingness to deception of outcome in a card game with binary outcome (win and loss)
Motor inhibitory control performance | before to after 7 nights of sleep restriction with and without acoustic stimulation
  inhibitory control performance measured by the stop-signal-task.
confidence | before to after 7 nights of sleep restriction with and without acoustic stimulation
  overconfidence measured by an incentivised procedure that elicits the certainity equivalent of a bet based on Performance in a quiz (cf. Murad et al. 2016 J Risk Uncertain)
overconfidence | before to after 7 nights of sleep restriction with and without acoustic stimulation
  overconfidence measured by an incentivised procedure that elicits the certainity equivalent of a bet based on Performance in a quiz (cf. Murad et al. 2016 J Risk Uncertain)
impulsivity | before to after 7 nights of sleep restriction with and without acoustic stimulation
  impulsivity as measured by an intertemporal choice Task.
Ocular inhibitory control performance | before to after 7 nights of sleep restriction with and without acoustic stimulation
  Ocular inhibitory control Performance measured by the Anti-Saccade Task.
Effort in inhibitory control performance | before to after 7 nights of sleep restriction with and without acoustic stimulation
  Pupil response (i.e. dilation) during a simple Go/No-Go Task.
Excessive daytime sleepiness | before to after 7 nights of sleep restriction with and without acoustic stimulation
  Excessive daytime sleepiness assessed by the Epworth sleepiness scale and the Stanford Sleepiness Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland